CLINICAL TRIAL: NCT02258269
Title: The Effect of Square Dance on Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Ph.D, Chengdu PLA General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SDRA00201401
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SQ (Experimental): Patients with rheumatoid arthritis exercise square dance
  Interventions: Other: SQ; Other: Control
- Control (Sham Comparator): Patients with rheumatoid arthritis listen to accompany music of square dance at home
  Interventions: Other: SQ; Other: Control

INTERVENTIONS:
Other: SQ
Other: Control

SUMMARY:
The purpose of this study is to observe the effect of square dance on rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* had wrist and/or MCP involvement
* aged 18 years diagnosed by rheumatology consultants with RA

Exclusion Criteria:

* severe psychological difficulties
* currently receiving mental health care
* any medical condition that might prevent them from safely exercising (e.g. history of more severe heart, lung or cerebrovascular disease)
* previously attended an education programme
* had a Modified Health Assessment Questionnaire score above 2 (0-3)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-08; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline Arthritis Helplessness Index (AHI) at 24 weeks | At 0 week, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Chengdu Military Area Command PLA, Chengdu, Sichuan, China